CLINICAL TRIAL: NCT02203422
Title: Recombinant Human Thrombopoietin (rhTPO) Combining Cyclosporin A Versus Cyclosporin A in Management of Steroid-Resistant/Relapsed Immune Thrombocytopenia （ITP）
Brief Title: A Multicenter Investigation of Recombinant Human Thrombopoietin (rhTPO) Combining Cyclosporin A Versus Cyclosporin A in Management of Steroid-Resistant/Relapsed Immune Thrombocytopenia （ITP）
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITP-Cyclosporin A
Record Dates: First submitted 2014-07-27; First posted 2014-07-29 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2014-07

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; Recombinant Human Thrombopoietin; Cyclosporin A
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination treatment group (Experimental): 60 enrolled patients are randomly picked up to take cyclosporin A in combination with rhTPO at the indicated dose.
  Interventions: Drug: Cyclosporin A; Drug: rhTPO
- single treatment group (Active Comparator): 60 enrolled patients are randomly picked up to take cyclosporin A at the indicated dose.
  Interventions: Drug: Cyclosporin A

INTERVENTIONS:
Drug: Cyclosporin A — given orally at a dose of 1.5-2.0mg/kg twice daily for 3 consecutive months, adjusted to maintain serum levels between 200-400 ng/ml and tapered by 50 mg/d per week if patients achieved a complete response.
Drug: rhTPO — given subcutaneously at a dose of 300 Units/kg for 14 consecutive days, following with a flexible dosage depending on platelet count until the 29th day
  Arms: combination treatment group

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other 5 well-known hospitals in China. In order to report the efficacy and safety of recombinant human thrombopoietin combining with cyclosporin A for the treatment of adults with refractory immune thrombocytopenia (ITP), compared to cyclosporin A monotherapy.

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of 120 steroid-resistant/relapsed ITP adult patients from 6 medical centers in China. One part of the participants are randomly selected to receive recombinant human thrombopoietin (given subcutaneously at a dose of 300 Units/kg for 14 consecutive days, following with a flexible dosage depending on platelet count until the 29th day), combining with cyclosporin A (given orally at a dose of 1.5-2.0mg/kg twice daily for 3 consecutive months, adjusted to maintain serum levels between 200-400 ng/ml and tapered by 50 mg/d per week if patients achieved a complete response). The others are selected to receive cyclosporin A monotherapy (given orally at a dose of 1.5-2.0mg/kg twice daily for 3 consecutive months, adjusted to maintain serum levels between 200-400 ng/ml and tapered by 50 mg/d per week if patients achieved a complete response). Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of the combination therapy compared to cyclosporin A monotherapy for the treatment of adults with steroid-resistant/relapsed ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Steroid-resistant/relapsed hospitalized patients, may be male or female, between the ages of 18-80 years.
3. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
4. Eastern Cooperative Oncology Group（ECOG）performance status ≤ 2.
5. Willing and able to sign written informed consent

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Current HIV infection or hepatitis B virus or hepatitis C virus infections. 3.Severe medical condition (lung, hepatic or renal disorder) other than ITP. 4.Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)

5.Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.

6.Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.

7.Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response (Complete Response) | The time frame is up to 3 months per subject
  CR. A complete response (CR) was defined as a sustained (≥ 3 months) platelet count ≥ 100×10^9/L
Evaluation of platelet response (Response) | The time frame is up to 3 months per subject
  R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia.
Evaluation of platelet response (No Response) | The time frame is up to 3 months per subject
  NR.No response (NR) was defined as platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.
Evaluation of platelet response (relapses) | The time frame is up to 3 months per subject
  A relapses was defined as platelet count falls below 30×10^9/L or bleeding accrues after achieving R or CR.

SECONDARY OUTCOMES:
The number and frequency of therapy associated adverse events The number and frequency of therapy associated adverse events The number and frequency of therapy associated adverse events The number and frequency of therapy associated adverse events | up to 3 months per subject

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr., Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China